CLINICAL TRIAL: NCT03171506
Title: Targeted Disruption to Cancer Metabolism Through Dietary Macronutrient Modification
Brief Title: Targeted Disruption to Cancer Metabolism and Growth Through Dietary Macronutrient Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Barbara Gower, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 317972
Record Dates: First submitted 2017-05-22; First posted 2017-05-31 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Ovarian Cancer; Endometrial Cancer
Keywords: ketogenic diet; carbohydrate-restricted diet
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms | interventions — Diet, Ketogenic; Diet

STUDY DESIGN:
Intervention Model Description: This study is a randomized clinical trial with a parallel arm design to evaluate the effects of 12 weeks of usual care plus AND or usual care plus KD on women with ovarian and endometrial cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care plus ketogenic diet (Experimental)
  Interventions: Other: Ketogenic diet
- Usual care plus AND diet (Placebo Comparator)
  Interventions: Other: AND diet

INTERVENTIONS:
Other: Ketogenic diet — Participants in the usual care plus ketogenic diet group will receive usual care plus dietary counseling in accordance with a ketogenic diet such that ~5% energy comes from carbohydrate, 25% energy from protein, and 70% energy from fat for the duration of the 12 week study.
  Arms: Usual care plus ketogenic diet
Other: AND diet — Participants in the usual care plus AND diet group will receive usual care plus dietary counseling in accordance with the Academy of Nutrition and Dietetics guidelines in 2013 for the duration of the 12 week study.
  Arms: Usual care plus AND diet

SUMMARY:
The objective of this investigation is to examine the effects of 12 weeks of usual care plus a ketogenic diet (KD) or usual care plus dietary recommendations endorsed by the Academy of Nutrition and Dietetics (AND) in women with ovarian and endometrial cancer. Participants undergo testing at baseline and at 12 weeks; the testing consists of blood draws, questionnaires, and measures of body composition. The baseline visit also includes a meeting with a registered dietitian to discuss the guidelines of the assigned diet.

It is hypothesized that the KD group will have improved cancer outcome measures, beneficial body composition changes, reduced fasting concentrations of glucose and insulin, and higher ratings of patient satisfaction with the diet relative to the AND group.

DETAILED DESCRIPTION:
This investigation is a randomized, controlled clinical trial among 66 (for a final n of 50) women with ovarian and endometrial cancer. Patients are randomized to one of two study arms for 12 weeks: usual care plus the ketogenic diet (KD) or usual care plus dietary recommendations endorsed by the Academy of Nutrition and Dietetics (AND).

Cases are accrued in the University of Alabama at Birmingham gynecologic oncology clinic. Patients are then randomized to one of the two diet groups using a blocked randomization strategy. The prescription for the AND follows the Academy's 2013 guidelines, with modifications as necessary of ovarian cancer. The KD has a macronutrient composition of ~5% energy from carbohydrate, 25% energy from protein, and 70% energy from fat. Carbohydrate foods include non-starchy vegetables (e.g., salad greens, green beans, summer squash). Patients are advised to avoid refined starches and added sugar and to emphasize consumption of whole foods. Protein foods include meat, poultry, fish, and eggs. Because protein can be converted to glucose in the liver via gluconeogenesis, patients are counseled to eat no more than ~100g protein per day, distributed across the day. Fat-containing foods include olive, coconut, and nut oils; butter; tree nuts and nut butters; cheese; cream; coconut milk; and avocados. Patients are counseled to obtain the majority of their fat intake from mono-unsaturated fatty acids (e.g., olive oil), and medium-chain triglycerides (e.g., coconut oil and milk); from nuts and nut butters; and from fresh fish. Full-fat dairy is limited to 4 ounces of cheese per day; butter is not limited. This diet is formulated to be low glycemic and anti-inflammatory, thereby lowering glucose, insulin, and markers of inflammation. Total energy intake is not restricted, as the focus is on insulin reduction rather than weight loss.

Diet interventions are provided by registered dietitians at the University of Alabama at Birmingham. Participants meet one-on-one with a dietitian at the baseline testing visit. Patients record food intake such that the dietitian can review them on a weekly basis, provide feedback, and tailor nutrition counseling; said counseling is delivered via phone and e-mail on a weekly basis throughout the 12-week intervention. Food records are analyzed for macronutrient composition, a range of micronutrients, and glycemic index.

Outcome measures include demographics (age, sex, race); body composition by dual X-ray absorptiometry (DXA) and bioelectrical impedance analysis (BIA); fasting concentrations of markers of inflammation, cancer progression (CA-125), and metabolism (glucose, insulin, ketones); cancer progression (as measured by CT scans done as part of usual care); quality of life (as measured by the Medical Outcomes Study Short Form-12 Health Survey, SF-12); satiety (as measured by a visual analog scale, VAS); and food cravings (as measured by the Food Craving Inventory, FCI).

Within groups changes in cancer markers, body composition, and other outcomes will be evaluated with paired t-tests. Between group differences will be evaluated with ANOVA/ANCOVA, controlling for relevant confounders (e.g., baseline values, age). Correlation analysis will be used to test the specific hypothesis that decrease in cancer outcomes across all patients will be associated with increase in serum ketone concentrations and decreasing concentration of fasting insulin. In a pilot study of 10 cancer patients, all of whom were placed on a KD, serum ketone production was increased to a greater extent (P<0.02) in those patients who showed remission or stable disease than in those patients who showed continued disease progression (Fine et al., 2012). Further, change in ketone production was associated with change in fasting insulin concentration. Thus, sample size calculations were based on change in fasting insulin using a previous diet intervention in a population of overweight/obese women with PCOS (Gower et al. 2013). In this study, a decrease in fasting insulin of 2.7 ± 4.6 µIU/ml was observed after 8 weeks of consumption of a eucaloric reduced-carbohydrate diet. Assuming a change of 2.7 ± 4.6 (µIU/ml), a two-sided paired t-test, and a significance alpha level of 0.05, we would have over 80% power to detect a significant change in fasting insulin with 25 participants per diet group. Allowing for 30% attrition, we plan to recruit 33 participants per diet group (total n=66).

Hypotheses include: 1) Cancer outcomes will improve in the KD group relative to the AND group, 2) The KD group will show a selective loss of visceral fat and preservation of lean mass, 3) Fasting concentrations of glucose, insulin, and insulin-like growth factor 1 (IGF-1) and its binding protein (IGFBP-1) will decline in the KD group but not in the AND group, 4) Changes in serum insulin concentration will be directly associated with changes in the cancer marker CA-125, 5) Changes in serum ketone concentration will be inversely associated with changes in cancer marker CA-125, and 6) Ratings of quality of life, food cravings, and satiety/hunger will improve in the KD group but not in the AND group.

ELIGIBILITY:
Inclusion Criteria:

* measurable disease or elevated CA-125
* classified as normal weight, overweight, or obese (BMI > 18.5)
* English speaking & reading
* can sign consent and are willing to be randomized and to adhere to the assigned protocol

Exclusion Criteria:

* pre-existing medical conditions that preclude enrollment: uncontrolled hypertension, myocardial infarction or cerebrovascular accident in the past six months, unstable angina within the last six months, congestive heart failure, serious infectious diseases, chronic hepatitis, cirrhosis, chronic malabsorption syndrome, chronic pancreatitis, chronic lung disease, major depressive or psychiatric disorder.
* current or medical condition that affects body weight such as uncontrolled hypo- or hyperthyroidism
* taking any of the following medications: anti-psychotic agents, monoamine oxidase inhibitors, antibiotics for HIV or tuberculosis, weight loss medications, or have taken weight loss medications in the last six months
* currently dieting

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This trial is limited to female participants, as it is a study of ovarian and endometrial cancer patients.
Enrollment: 57 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-07-18 (Actual)

PRIMARY OUTCOMES:
change in fasting glucose | 12 weeks
  mg/dL
change in fasting insulin | 12 weeks
  uU/mL
change in fasting beta-hydroxybutyrate | 12 weeks
  mM

SECONDARY OUTCOMES:
CA-125 | baseline and 12 weeks
  U/mL
IGF-1 | baseline and 12 weeks
  ng/mL
IGFBP-1 | baseline and 12 weeks
  ug/mL
markers of inflammation | baseline and 12 weeks
  fasting serum concentrations of a variety of inflammatory markers
total body fat | baseline and 12 weeks
  g, measured by DXA and BIA
regional body fat | baseline and 12 weeks
  g, measured by DXA and BIA
total lean mass | baseline and 12 weeks
  g, measured by DXA and BIA
regional lean mass | baseline and 12 weeks
  g, measured by DXA and BIA
quality of life | baseline and 12 weeks
  Physical and mental health functioning as assessed by the Medical outcomes Study Short Form-12 Health Survey, which produces a physical component summary and mental component summary score.
perceived hunger | baseline and 12 weeks
  Perceived hunger assessed by a visual analog scale
food cravings | baseline and 12 weeks
  Cravings for particular types foods (fats, sweets, starches) as assessed by the Food Craving Inventory
lipids | baseline and 12 weeks
  fasting serum concentrations of total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Gower, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gower BA, Chandler-Laney PC, Ovalle F, Goree LL, Azziz R, Desmond RA, Granger WM, Goss AM, Bates GW. Favourable metabolic effects of a eucaloric lower-carbohydrate diet in women with PCOS. Clin Endocrinol (Oxf). 2013 Oct;79(4):550-7. doi: 10.1111/cen.12175. Epub 2013 May 20. PMID 23444983
- [Background] Fine EJ, Segal-Isaacson CJ, Feinman RD, Herszkopf S, Romano MC, Tomuta N, Bontempo AF, Negassa A, Sparano JA. Targeting insulin inhibition as a metabolic therapy in advanced cancer: a pilot safety and feasibility dietary trial in 10 patients. Nutrition. 2012 Oct;28(10):1028-35. doi: 10.1016/j.nut.2012.05.001. Epub 2012 Jul 26. PMID 22840388
- [Derived] Cohen CW, Fontaine KR, Arend RC, Soleymani T, Gower BA. Favorable Effects of a Ketogenic Diet on Physical Function, Perceived Energy, and Food Cravings in Women with Ovarian or Endometrial Cancer: A Randomized, Controlled Trial. Nutrients. 2018 Aug 30;10(9):1187. doi: 10.3390/nu10091187. PMID 30200193
- [Derived] Cohen CW, Fontaine KR, Arend RC, Alvarez RD, Leath CA III, Huh WK, Bevis KS, Kim KH, Straughn JM Jr, Gower BA. A Ketogenic Diet Reduces Central Obesity and Serum Insulin in Women with Ovarian or Endometrial Cancer. J Nutr. 2018 Aug 1;148(8):1253-1260. doi: 10.1093/jn/nxy119. PMID 30137481